CLINICAL TRIAL: NCT03072160
Title: Phase II Trial of Pembrolizumab in Recurrent or Metastatic Medullary Thyroid Cancer
Brief Title: Pembrolizumab in Recurrent or Metastatic Medullary Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ravi A. Madan, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170061; 17-C-0061
Record Dates: First submitted 2017-03-03; First posted 2017-03-07 (Actual); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Medullary Thyroid Cancer (MTC)
Keywords: Anti-PD1/PDL1; Vaccine Therapy; TKI-Naive
MeSH Terms: conditions — Carcinoma, Medullary | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort 1: Participants that had an immune stimulating cancer vaccine (Experimental): Pembrolizumab 200 mg will be administered as a 30 minute intravenous (IV) infusion every 3 weeks for two years.
  Group 1: cancer vaccine
  Interventions: Drug: Pembrolizumab
- Cohort 2: Participants that have had no vaccine (Experimental): Pembrolizumab 200 mg will be administered as a 30 minute intravenous (IV) infusion every 3 weeks for two years.
  Group 2: had no previous vaccine
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg will be administered as a 30 minute intravenous (IV) infusion every 3 weeks.
  Other Names: Lambrolizumab; MK-3475

SUMMARY:
Background:

Medullary thyroid cancer (MTC) is a tumor of the thyroid gland. Surgery is the only current treatment to cure it. The drug pembrolizumab (MK-3475) is a new type of cancer therapy. It works by allowing the immune system to detect and kill tumor cells.

Objective:

To test how pembrolizumab affects people with MTC and if it can offer them clinical benefit.

Eligibility:

People ages 18 and older with MTC

Patients who have recurrent or metastatic MTC, for whom surgery is not a curative option

Patients with some imaging evidence of MTC

Patients with minimal symptoms related to MTC

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Blood, urine, and heart tests
* Computed tomography (CT) scan or magnetic resonance imaging (MRI): They lie in a machine that takes pictures of the body.
* Bone scan

Participants will be put in a group based on their treatment history:

* Group 1 if they have had an immune stimulating cancer vaccine
* Group 2 if they have had no vaccine

Participants will receive the study drug as a 30-minute intravenous (IV) infusion every 3 weeks. Treatment will continue for up to 2 years as long as they tolerate it and their disease does not get worse.

Participants will have physical exams and blood tests on the day of each infusion. They will have CT and bone scans every 3 months.

Participants may save biopsies before treatment and after starting treatment.

Participants will have a final visit 3-4 weeks after stopping treatment. This will include a physical exam and blood and heart tests.

After this study, participants can join a long-term follow-up study.

DETAILED DESCRIPTION:
Background:

* Anti-programmed cell death protein 1 (PD1)/programmed death-ligand 1 (PDL1) therapies have had clinical success in a minority of unselected patients across multiple tumor types
* While many questions remain about optimal PD1/PDL1 staining techniques to pre-select responders, less focus is being place on how to optimize responses in a broader cohort of patients
* Emerging preclinical and clinical data supports the hypothesis that a strong immunologic response in the tumor microenvironment induces PDL1 expression on the tumor and is associated with better clinical response to anti-PD1/PDL1 therapies
* Therapeutic cancer vaccines are one strategy to induce an immunologic response to the tumor, thereby enhancing PDL1 expression and optimizing clinical responses across all patients
* Limited clinical data exists about the potential benefit of sequential therapy with a therapeutic cancer vaccine followed by PD1/PDL1 inhibition
* This study will explore the role of PD1 inhibition in medullary thyroid cancer and evaluate the potential differences based on previous vaccine therapy

Objective:

-The primary objective of this trial is to determine whether administering a PD1 inhibitor to patients with medullary thyroid cancer will permit a modest fraction to be able to experience a 50% or greater decline in calcitonin levels or experience a partial/complete response on imaging

Key Eligibility:

* Patients greater than or equal to 18 years of age with evidence of metastatic medullary thyroid cancer including disease that is evaluable on bone, computed tomography (CT) scan or magnetic resonance imaging (MRI)
* Must have elevated calcitonin levels greater than 40 pg/mL
* Patients with minimal or no disease related-symptoms (minimal symptoms will include those that do not affect activities of daily living or pain that does not require regularly schedule narcotics)
* Eastern Cooperative Oncology Group (ECOG) 0-1
* Should have no autoimmune diseases; no evidence of being immunocompromised; no serious inter-current medical illness
* No brain metastasis, history of seizures, encephalitis, or multiple sclerosis

Design:

* This is a phase II, open label, single center clinical trial where all patients receive the anti-PD1/PDL1 therapy pembrolizumab
* Patients will enroll in one of two cohorts: patients with previous vaccine therapy or patients without previous vaccine therapy
* All patients will be TKI naive with minimal symptoms (consistent with the eligibility for our current study)
* Based on our calcitonin findings with our current study of 30 patients, we have determined that a confirmed calcitonin decline of 50% would be a rare finding, providing compelling preliminary evidence of clinical activity
* A total of 30 patients will be enrolled in the proposed study (15 patients in each cohort). Given that we already have 30 patients on a study with vaccine, we would only need to identify and recruit 15 patients for the vaccine-naive cohort.
* Based on these metrics, we could have >6 months of calcitonin data in 30 patients within 2 years from trial initiation
* Additional immune correlative capitalizing on the extensive immune monitoring experience of the Laboratory of Tumor Immunology and Biology (LTIB) will allow for assessments of antigen specific T-cells and 123 immune subsets. These findings could provide the basis for biomarker development when taken together with biochemical and clinical responses seen in this study

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis: Patients must have histologically confirmed medullary thyroid cancer by the Laboratory of Pathology or a pathology report and history consistent with medullary thyroid cancer. It is not uncommon for a secondary, minor pathologic focus of another form of thyroid cancer to be coincidentally found in 15-20% of patients with medullary thyroid cancer. In such cases, eligibility is based on the discretion of the investigator.
* Patients must have evidence of metastatic medullary thyroid cancer including disease that is evaluable on bone, computed tomography (CT) scan or magnetic resonance imaging (MRI). (Patients who are surgical candidates and potentially rendered disease free with surgical resection are not eligible.)
* Patients must have elevated calcitonin levels greater than 40 pg/mL
* Patients must have minimal or no disease related-symptoms (Minimal symptoms will include those that do not affect activities of daily living or pain that does not require regularly scheduled narcotics.)
* Patients must have evaluable disease on imaging
* No history of seizures, encephalitis, or multiple sclerosis.
* Age greater than or equal to 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 at study entry (Karnofsky greater than or equal to 70).
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception, Contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception. Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Willing to travel to the National Institutes of Health (NIH) for follow-up visits
* Able to understand and sign informed consent.
* Demonstrate adequate organ function, all screening labs should be performed within 10 days of treatment initiation.
* Adequate Organ Function Laboratory Values

  * Hematological

    ---Absolute neutrophil count (ANC) greater than or equal to1,000 /mcL
  * Platelets greater than or equal to 100,000 / mcL
  * Hemoglobin greater than or equal to 9 g/dL or greater than or equal to 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
  * Renal

    * Serum creatinine less than or equal to1.5 X upper limit of normal (ULN) OR
    * Measured or calculated* creatinine clearance (Glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl) greater than or equal to 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
  * Hepatic

    * Serum total bilirubin less than or equal to 1.5 X ULN OR Direct bilirubin less than or equal to ULN for subjects with total bilirubin levels > 1.5 ULN
    * Aspartate aminotransferase (AST) Serum glutamic-oxaloacetic transaminase (SGOT) and Alanine aminotransferase (ALT) Serum glutamic pyruvic transaminase (SGPT) less than or equal to 2.5 X ULN OR less than or equal to 5 X ULN for subjects with liver metastases
    * Albumin >2.5 mg/dL
  * Coagulation

    * International Normalized Ratio (INR) or Prothrombin Time (PT) less than or equal to1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
    * Activated Partial Thromboplastin Time (aPTT) less than or equal to1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

      * Creatinine clearance should be calculated per Cockcroft-Gault equation

EXCLUSION CRITERIA:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had prior targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., less than or equal to Grade 1 or at baseline) from adverse events due to a previously administered agent. Note: Subjects with less than or equal to Grade 2 neuropathy are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable for 6 months (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subjects participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breast feeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-Programmed cell death protein 1 (PD-1), anti- programmed cell death-1 ligand 1 (PD-L1), or anti-Programmed death ligand 2 (PD-L2) agent.
* Has Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., hepatitis C virus (HCV) ribonucleic acid (RNA) [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy
* Concurrent use of systemic steroids, except for physiologic doses of systemic steroid replacement or local (topical, nasal, eye drops or inhaled) steroid use. Limited doses of systemic steroids (e.g., in patients with exacerbations of reactive airway disease or to prevent intravenous (IV) contrast allergic reaction or anaphylaxis in patients who have known contrast allergies) are allowed.
* Serious inter-current medical illness which would interfere with the ability of the patient to carry out the treatment program.
* Patients with second malignancy within 3 years of enrollment; Patients curatively treated non-melanoma skin cancers or carcinoma in situ of the bladder, are not excluded. Patients with Multiple endocrine neoplasia type 2 (MEN2) and a history of pheochromocytoma will also not be excluded. In addition, patients with prostate cancer who do not require systemic therapy will not be excluded. (A secondary, minor pathologic focus of another form of thyroid cancer may be coincidentally found in 15-20% of patients with medullary thyroid cancer. In such cases, eligibility is based on the discretion of the investigator.)
* Patients with previous history of vandetanib or cabozantinib treatment for more than 28 days of treatment (patients have discontinued treatment for 28 days before enrolling).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-06-16 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi A Madan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-C-0061.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Cancer Vaccine: Pembrolizumab 200 mg will be administered as a 30 minute intravenous (IV) infusion every 3 weeks for two years.
  Group 1: cancer vaccine
  Pembrolizumab: Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks.
- Cohort 2: Participants That Have Had No Vaccine: Pembrolizumab 200 mg will be administered as a 30 minute intravenous (IV) infusion every 3 weeks for two years.
  Group 2: had no previous vaccine
  Pembrolizumab: Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks.
Period: Overall Study
Arm/Group | Cohort 1: Cancer Vaccine | Cohort 2: Participants That Have Had No Vaccine
Started | 13 | 4
Completed | 2 | 0
Not Completed | 11 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Refused further treatment | 6 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Disease progression on study | 1 | 1
Not completed — No contact | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Cancer Vaccine | Cohort 2: Participants That Have Had No Vaccine | Total
Number analyzed (Participants) | 13 | 4 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 2 | 12
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.82 (11.8) | 59.48 (11.85) | 56.15 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 3 | 13
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 3 | 14
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 9 | 4 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 4 | 17
Median Baseline Carcinoembryonic Antigen (CEA) [Median (Full Range); unit: ng/ml] — Normal level is <2.5ng/ml. A large magnitude decline in CEA may be associated with tumor responses.
  ng/ml | 125 [3.7 to 1650] | 207 [153 to 943] | 175 [3.7 to 1650]
Median Baseline Calcitonin [Median (Full Range); unit: pg/ml] — Normal level is <10pg/ml. A large magnitude decline in calcitonin may be associated with tumor responses.
  pg/ml | 509 [65 to 35,607] | 6000 [2672 to 103,312] | 6000 [65 to 103,312]

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response
Description: Participants with medullary thyroid cancer were administered a programmed cell death protein 1 (PD1) inhibitor to determine if any experienced a 50% or greater decline in calcitonin levels. A calcitonin response is defined as participants with a ≥50% decline from baseline that is then confirmed on a subsequent calcitonin assessment at least one week later.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Cancer Vaccine | Cohort 2: Participants That Have Had No Vaccine
Number analyzed (Participants) | 13 | 4
Participants | 0 | 0

2. Primary Outcome: Percentage of Participants With a Partial Response and Complete Response by Computed Tomography (CT) or Magnetic Resonance Imaging (MRI)
Description: Participants were imaged by CT or MRI and followed for response using the Immune-Related Response Criteria (irRC). Partial Response is a ≥30% decrease in the sum of the largest diameter (SLD) compared with baseline confirmed by a consecutive assessment at least 4 weeks after the first documentation. Complete Response is a 100% disappearance of all lesions, whether measurable or not, and no new lesions, in two consecutive observations not less than 4 weeks from the date first documented.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Cancer Vaccine | Cohort 2: Participants That Have Had No Vaccine
Number analyzed (Participants) | 13 | 4
Participants | 0 | 0

3. Secondary Outcome: Percentage Change in (Cluster of Differentiation 4 (CD4), CD8, Tregs, and Natural Killer (NK) Cells at Day 1 and 84 Days in All Participants
Description: Regulatory T-Cells (CD4, CD8, Tregs, and NK cells) in peripheral blood mononuclear cell (PBMC)s were measured by 7-color flow cytometry.
Time Frame: Day 1 and 84 days
Measure: Mean (Full Range); unit: Percentage change
Groups:
- All Participants at Day 1; All Participants at Day 84: All participants in group 1 and group 2.
  Group 1: cancer vaccine
  Group 2: had no previous vaccine
Arm/Group | All Participants at Day 1 | All Participants at Day 84
Number analyzed (Participants) | 16 | 16
Percentage change
  CD4 | 34.73 [12.5 to 53.5] | 33.95 [9.7 to 46.5]
  CD8 | 13.70 [6.17 to 26.3] | 12.50 [6.5 to 24.22]
  Tregs | 0.70 [0.0 to 1.2] | 0.77 [0.46 to 1.8]
  NK | 10.47 [6.6 to 17.7] | 10.26 [4.6 to 19.5]
Statistical Analysis 1: Comparison: All Participants at Day 1 vs All Participants at Day 84; Test type: Other; p = 0.926, Wilcoxon signed-rank test — CD4; A change is defined as being statistically significant (p>0.05)
Statistical Analysis 2: Comparison: All Participants at Day 1 vs All Participants at Day 84; Test type: Other; p = 0.445, Wilcoxon signed-rank test — CD8; A change is defined as being statistically significant (p>0.05)
Statistical Analysis 3: Comparison: All Participants at Day 1 vs All Participants at Day 84; Test type: Other; p = 0.210, Wilcoxon signed-rank test — Tregs; A change is defined as being statistically significant (p>0.05)
Statistical Analysis 4: Comparison: All Participants at Day 1 vs All Participants at Day 84; Test type: Other; p = 0.780, Wilcoxon signed-rank test — Natural Killer (NK) cells; A change is defined as being statistically significant (p>0.05)

4. Secondary Outcome: Number of Participants With a Sustained Decline in Carcinoembryonic Antigen (CEA)
Description: A sustained 50% decline in CEA. A large magnitude decline in CEA may be associated with tumor responses.
Time Frame: every 3 weeks while on treatment and post treatment, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Cancer Vaccine | Cohort 2: Participants That Have Had No Vaccine
Number analyzed (Participants) | 13 | 4
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With a Sustained Decline in Calcitonin
Description: A sustained 50% decline in calcitonin. A large magnitude decline in calcitonin may be associated with tumor responses.
Time Frame: every 3 weeks while on treatment and post treatment, up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Cancer Vaccine | Cohort 2: Participants That Have Had No Vaccine
Number analyzed (Participants) | 13 | 4
Participants | 0 | 0

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression, assessed by the Immune-Related Response Criteria (irRC), is defined as at least 20% increase in the sum of the largest diameter (SLD) compared with nadir (minimum recorded tumor burden) and an increase of at least 5mm over the nadir, confirmed by a repeat,consecutive observations at least 4 weeks from the date first documented.
Time Frame: 3 weeks for up to 2 years while on treatment than 2 weeks after last treatment
Measure: Number; unit: Days
Arm/Group | Cohort 1: Cancer Vaccine | Cohort 2: Participants That Have Had No Vaccine
Number analyzed (Participants) | 1 | 1
Days | 210 | 55

7. Secondary Outcome: Overall Survival at 2 Years
Description: Percentage of participants who are alive at 2 years.
Time Frame: 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: Cancer Vaccine | Cohort 2: Participants That Have Had No Vaccine
Number analyzed (Participants) | 13 | 4
percentage of participants | 100 | 50

8. Secondary Outcome: Number of Participants With Grade ≥1 Adverse Events Possibly, Probably, or Definitely Related to Pembrolizumab
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe or medically significant but not immediately life-threatening. Grade 4 is life-threatening; urgent intervention indicated. Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately 25 months and 28 days for cohort 1 and 18 months and 12 days for cohort 2.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Grade 1 Possibly Related; Cohort 1: Grade 2 Possibly Related; Cohort 1: Grade 3 Possibly Related; Cohort 2: Grade 1 Possibly Related; Cohort 2: Grade 2 Possibly Related; Cohort 2: Grade 3 Possibly Related: Adverse events possibly related to Pembrolizumab.
- Cohort 1: Grade 1 Probably Related; Cohort 1: Grade 2 Probably Related; Cohort 1: Grade 3 Probably Related; Cohort 2: Grade 1 Probably Related; Cohort 2: Grade 2 Probably Related; Cohort 2: Grade 3 Probably Related: Adverse events probably related to Pembrolizumab.
- Cohort 1: Grade 1 Definitely Related; Cohort 1: Grade 2 Definitely Related; Cohort 1: Grade 3 Definitely Related; Cohort 2: Grade 1 Definitely Related; Cohort 2: Grade 2 Definitely Related; Cohort 2: Grade 3 Definitely Related: Adverse events definitely related to Pembrolizumab.
Arm/Group | Cohort 1: Grade 1 Possibly Related | Cohort 1: Grade 1 Probably Related | Cohort 1: Grade 1 Definitely Related | Cohort 1: Grade 2 Possibly Related | Cohort 1: Grade 2 Probably Related | Cohort 1: Grade 2 Definitely Related | Cohort 1: Grade 3 Possibly Related | Cohort 1: Grade 3 Probably Related | Cohort 1: Grade 3 Definitely Related | Cohort 2: Grade 1 Possibly Related | Cohort 2: Grade 1 Probably Related | Cohort 2: Grade 1 Definitely Related | Cohort 2: Grade 2 Possibly Related | Cohort 2: Grade 2 Probably Related | Cohort 2: Grade 2 Definitely Related | Cohort 2: Grade 3 Possibly Related | Cohort 2: Grade 3 Probably Related | Cohort 2: Grade 3 Definitely Related
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 13 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4
Participants
  Acute kidney injury | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Allergic rhinitis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anorexia | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diarrhea | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dizziness | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dry eye | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dry skin | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eye disorders | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eye pain | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue | 6 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Flashing lights | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Flu-like symptoms | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Generalized muscle weakness | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Headache | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hearing impaired | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Injection site reaction | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Nausea | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil count decreased | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain in extremity | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain of skin | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet count decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pruritis | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash acneiform | 4 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash maculopapular | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Renal and urinary disorders | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin and subcutaneous tissue disorders | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Grade ≥1 Adverse Events Unlikely or Unrelated to Pembrolizumab
Description: as for outcome 8
Time Frame: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Grade 1 Unlikely Related; Cohort 1: Grade 2 Unlikely Related; Cohort 1: Grade 3 Unlikely Related; Cohort 2: Grade 1 Unlikely Related; Cohort 2: Grade 2 Unlikely Related; Cohort 2: Grade 3 Unlikely Related: Adverse events unlikely related to Pembrolizumab.
- Cohort 1: Grade 1 Unrelated; Cohort 1: Grade 2 Unrelated; Cohort 1: Grade 3 Unrelated; Cohort 2: Grade 1 Unrelated; Cohort 2: Grade 2 Unrelated; Cohort 2: Grade 3 Unrelated: Adverse events unrelated to Pembrolizumab.
Arm/Group | Cohort 1: Grade 1 Unlikely Related | Cohort 1: Grade 1 Unrelated | Cohort 1: Grade 2 Unlikely Related | Cohort 1: Grade 2 Unrelated | Cohort 1: Grade 3 Unlikely Related | Cohort 1: Grade 3 Unrelated | Cohort 2: Grade 1 Unlikely Related | Cohort 2: Grade 1 Unrelated | Cohort 2: Grade 2 Unlikely Related | Cohort 2: Grade 2 Unrelated | Cohort 2: Grade 3 Unlikely Related | Cohort 2: Grade 3 Unrelated
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13 | 13 | 4 | 4 | 4 | 4 | 4 | 4
Participants
  Abdominal pain | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Alanine aminotransferase increased | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Allergic rhinitis | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Anemia | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Anorexia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Aspartate aminotransferase increased | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Back pain | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood bilirubin increased | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Buttock pain | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cataract | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Cough | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CPK increased | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dehydration | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Diarrhea | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Dizziness | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dry mouth | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dry skin | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Dyspnea | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Ear and labyrinth disorders | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema face | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Edema limbs | 0 | 2 | 00 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Enterocolitis | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eye disorders | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Eye pain | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Fatigue | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Flank pain | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Flushing | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 00 | 0 | 0 | 0
  Gait disturbance | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  General disorders & admin. site conditions | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Generalized muscle weakness | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Headache | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperglycemia | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Hypoalbuminemia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia | 0 | 8 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
  Hypokalemia | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hyponatremia | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Insomnia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lip pain | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte count decreased | 0 | 4 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Menopause | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nail ridging | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Nasal congestion | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Nausea | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Neck pain | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain | 0 | 6 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pain in extremity | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White blood cell decreased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increased | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  Hyperuricemia | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Upper respiratory infection | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Peripheral motor neuropathy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Respiratory, thoracic and mediastinal disorders | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypotension | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Presyncope | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Wheezing | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Skin infection | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Paresthesia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rhinitis infective | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash acneiform | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Cancer Vaccine | Cohort 2: Participants That Have Had No Vaccine
Number analyzed (Participants) | 13 | 4
Participants | 13 | 4

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 25 months and 28 days for cohort 1 and 18 months and 12 days for cohort 2.
Groups:
- Cohort 1: Cancer Vaccine: Pembrolizumab 200 mg will be administered as a 30 minute intravenous (IV) infusion every 3 weeks for two years.
  Group 1: had an immune stimulating cancer vaccine previously
  Pembrolizumab: Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks.
Arm/Group | Cohort 1: Cancer Vaccine | Cohort 2: Participants That Have Had No Vaccine
All-Cause Mortality (participants affected / at risk) | 0/13 | 2/4
Serious Adverse Events (participants affected / at risk) | 2/13 | 2/4
Other Adverse Events (participants affected / at risk) | 13/13 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Cancer Vaccine (N=13) | Cohort 2: Participants That Have Had No Vaccine (N=4)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, Acute interstitial nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Cancer Vaccine (N=13) | Cohort 2: Participants That Have Had No Vaccine (N=4)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (7) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
CPK increased (Investigations) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Creatinine increased (Investigations) | 2 (7) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 4 (8) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ear and labyrinth disorders - Other, ear clogged (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, tugging / fluid (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 2 (2) | 1 (1)
Enterocolitis (Infections and infestations) | 1 (1) | 0 (0)
Eye disorders - Other, Itching eyes (both eyes) (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, L eye swelling (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, redness right eye (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other, Blepharitis, eye tearing and mild blurry vision (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, Eye fullness (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 2 (3) | 0 (0)
Fatigue (General disorders) | 6 (8) | 3 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flashing lights (Eye disorders) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, lightheadedness transient (General disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (6) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (7) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 9 (20) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 3 (10) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 4 (5) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (11) | 2 (4)
Menopause (Social circumstances) | 1 (1) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (5) | 0 (0)
Pain (General disorders) | 6 (9) | 1 (1)
Pain in extremity (General disorders) | 4 (4) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 (11) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Intermittent skin itching, Comes and goes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Itching intermittently after shower (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 3 (4) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT03072160/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT03072160/ICF_001.pdf